CLINICAL TRIAL: NCT00813956
Title: A Phase 2 Study of Standard Chemotherapy Plus BSI-201 (a PARP Inhibitor) in the Neoadjuvant Treatment of Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11487; 20080206 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: triple negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Gemcitabine; Carboplatin; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): standard chemotherapy plus BSI-201
  Interventions: Drug: gemcitabine plus carboplatin plus BSI-201

INTERVENTIONS:
Drug: gemcitabine plus carboplatin plus BSI-201 — iv, 3 week cycles

SUMMARY:
This study will investigate whether the neoadjuvant combination of gemcitabine, carboplatin, and BSI-201 will cause a high percentage of triple negative breast cancer patients to achieve a pathologic complete response prior to surgery.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer
* stage I-IIIA disease
* ER, PR, Her2/neu-negative status
* no prior treatment for breast cancer
* age 18 years of greater
* normal renal, liver function
* normal hematologic status
* ECOG Performance status 0, 1
* Evaluation by a surgeon to determine breast conservation eligibility
* Women of childbearing potential must have a documented negative pregnancy test within 2 months of study trial entry and agree to birth control during the duration of the trial therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Metastatic breast cancer
* Inoperable breast cancer, including Stage IIIB and IIIC
* Tumor size less than 1 centimeter
* Prior surgery, systemic therapy, or radiotherapy for the current cancer
* Hormone receptor-positive breast cancer
* Her2/neu-positive breast cancer
* Any concurrent condition which in the investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Pregnant or nursing women
* Receipt of any investigational agents within 30 days prior to commencing study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
pathologic complete response | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Stanford Comprehensive Cancer Center, Stanford, California
  - PrECOG, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Telli ML, Jensen KC, Vinayak S, Kurian AW, Lipson JA, Flaherty PJ, Timms K, Abkevich V, Schackmann EA, Wapnir IL, Carlson RW, Chang PJ, Sparano JA, Head B, Goldstein LJ, Haley B, Dakhil SR, Reid JE, Hartman AR, Manola J, Ford JM. Phase II Study of Gemcitabine, Carboplatin, and Iniparib As Neoadjuvant Therapy for Triple-Negative and BRCA1/2 Mutation-Associated Breast Cancer With Assessment of a Tumor-Based Measure of Genomic Instability: PrECOG 0105. J Clin Oncol. 2015 Jun 10;33(17):1895-901. doi: 10.1200/JCO.2014.57.0085. Epub 2015 Apr 6. PMID 25847929